CLINICAL TRIAL: NCT00489359
Title: A Phase 1 and 2 Clinical Trial of ALIMTA® (Pemetrexed) in Combination With Carboplatin in Patients With Recurrent Ovarian or Primary Peritoneal Cancer
Brief Title: Trial of Pemetrexed and Carboplatin in Patients With Recurrent Ovarian or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9516; H3E-MC-JMHH (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Results first posted 2011-06-16 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-05

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed/Carboplatin Phase 1 (Experimental): Pemetrexed was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle.
  Carboplatin was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion.
  Interventions: Drug: Pemetrexed - Phase 1; Drug: Carboplatin - Phase 1
- Pemetrexed/Carboplatin Phase 2 (Experimental): Pemetrexed was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle.
  Carboplatin was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion.
  Interventions: Drug: Pemetrexed - Phase 2; Drug: Carboplatin - Phase 2

INTERVENTIONS:
Drug: Pemetrexed - Phase 1 — 500, 600, 700, 800, or 900 milligrams per square meter (mg/m^2), administered intravenously (IV), every 21 days x 6 cycles, dose escalate to Maximum Tolerated Dose (MTD)
  Other Names: LY231514; Alimta
  Arms: Pemetrexed/Carboplatin Phase 1
Drug: Carboplatin - Phase 1 — area under the concentration time curve (AUC) 5 or 6 mg/mL*min, administered intravenously (IV), every 21 days x 6 cycles, dose escalation to Maximum Tolerated Dose (MTD)
  Arms: Pemetrexed/Carboplatin Phase 1
Drug: Pemetrexed - Phase 2 — Dose determined from Phase 1: 500 mg/m^2, administered IV, every 21 days x 6 cycles
  Other Names: LY231514; Alimta
  Arms: Pemetrexed/Carboplatin Phase 2
Drug: Carboplatin - Phase 2 — Dose determined from Phase 1: AUC 6 mg/mL*min, administered IV, every 21 days x 6 cycles
  Arms: Pemetrexed/Carboplatin Phase 2

SUMMARY:
The purpose of this study is to determine efficacy of the combination therapy of pemetrexed and carboplatin as treatment for patients with platinum-sensitive ovarian cancer. This study also includes patients with primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ovarian or primary peritoneal cancer confirmed by pathology
* Patients must have recurrent ovarian cancer which is sensitive to platinum therapy
* Prior radiation therapy is allowed

Measurable disease as defined by the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines, or non-measurable but cancer antigen 125 (CA-125) greater than or equal to 2X upper limit.

Exclusion Criteria:

* More than 2 lines of therapy for ovarian or primary peritoneal cancer.
* Pregnant or breast feeding.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bahía Blanca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ramos Mejía
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salta
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
- Germany (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bonn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chemnitz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Düsseldorf
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
- Poland (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olsztyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Sweden (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gothenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lund

REFERENCES:
- [Background] Bookman MA. 2006. GOG0182-ICON5: 5-arm phase III randomized trial of paclitaxel (P) and carboplatin (C) vs combinations with gemcitabine (G), PEG-lipososomal doxorubicin (D), or topotecan (T) in patients (pts) with advanced-stage epithelial ovarian (EOC) or primary peritoneal (PPC) carcinoma. J Clin Oncol 24 (suppl 18S). Abstract 5002.
- [Derived] Sehouli J, Alvarez AM, Manouchehrpour S, Ghatage P, Szczylik C, Zimmermann A, Bauknecht T, Look KY, Oskay-Oezcelik G. A phase II trial of pemetrexed in combination with carboplatin in patients with recurrent ovarian or primary peritoneal cancer. Gynecol Oncol. 2012 Feb;124(2):205-9. doi: 10.1016/j.ygyno.2011.09.007. Epub 2011 Nov 1. PMID 22044606
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase 1 and Phase 2 were conducted in different participants (i.e., Phase 1 participants did not also participate in Phase 2).
Groups:
- Pemetrexed/Carboplatin Phase 1: Pemetrexed (500, 600, 700, 800, or 900 mg/m^2) was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle. Carboplatin [area under the concentration-time curve (AUC) 5 or 6 mg/mL*min] was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion. Participant accrual and dose escalations were dependent upon the observed pattern of dose limiting toxicity (DLT). If none of the 3 initial participants of a given dose level experienced a DLT in Cycle 1, enrollment proceeded to the next dose level.
- Pemetrexed/Carboplatin Phase 2: Pemetrexed (500 mg/m^2) was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle. Carboplatin (AUC 6 mg/mL*min) was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion.
Period: Overall Study
Arm/Group | Pemetrexed/Carboplatin Phase 1 | Pemetrexed/Carboplatin Phase 2
Started | 20 | 66
Completed | 13 (Received at least 6 cycles of therapy. Not completed implies participant received <6 cycles.) | 37 (Received at least 6 cycles of therapy. Not completed implies participant received <6 cycles.)
Not Completed | 7 | 29
Not completed — Death | 0 | 2
Not completed — Progressive Disease | 5 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Adverse Event | 0 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed/Carboplatin Phase 1 | Pemetrexed/Carboplatin Phase 2 | Total
Number analyzed (Participants) | 20 | 66 | 86
Age Continuous [Mean (Standard Deviation); unit: years] | 56.99 (11.06) | 57.71 (10.44) | 57.54 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 66 | 86
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 20 | 59 | 79
  Hispanic | 0 | 7 | 7
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 7 | 7
  Argentina | 0 | 14 | 14
  Poland | 0 | 5 | 5
  Germany | 20 | 31 | 51
  Sweden | 0 | 9 | 9
Performance Status [Number; unit: participants] — The Eastern Cooperative Oncology Group (ECOG) score is an overall assessment of the functional/physical performance of the patient. Scores are:
  0=Fully active, able to carry on all pre-disease performance without restriction. 1=Restricted in strenuous activity but ambulatory and able to carry out work of a sedentary nature. 2=Ambulatory and capable of self care but unable to carry out any work activities: up and about more than 50% of time. 3=Capable of only limited self care, confined to bed or chair more than 50% of waking hours. 4=Completely disabled, cannot carry on any self care.
  participants
    ECOG Status 0 | 3 | 46 | 49
    ECOG Status 1 | 17 | 20 | 37
Tumor Type [Number; unit: participants]
  Ovarian Cancer | 15 | 61 | 76
  Peritoneal Cancer | 5 | 5 | 10
Platinum-free interval [Number; unit: participants] — The time elapsed since completing platinum-based therapy.
  participants
    <6 months | 0 | 3 | 3
    6-12 months | 6 | 23 | 29
    >12 months | 14 | 40 | 54

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - Maximum Tolerated Dose (MTD) of Pemetrexed in Combination With Carboplatin
Description: MTD was to be determined by increasing doses of pemetrexed up to 900 mg/m^2 and carboplatin Area Under the Concentration-Time Curve (AUC) up to 6 mg/mL*min based on observed pattern of dose limiting toxicity (DLT). See Outcome #3 for DLT. If none of 3 initial participants at a given level experienced a DLT in Cycle 1, enrollment proceeded to the next dose level. If at least 2 participants experienced a DLT in Cycle 1 at a dose level, that dose level was considered the MTD. However, based on results from a different Phase 2 Study (NCT00109096), further dose escalations were not explored.
Time Frame: First treatment to toxicity (up to 18 months)
Population: MTD was not determined in this study, so zero participants were analyzed.
Measure: Number; unit: mg/m^2
Groups:
- Pemetrexed/Carboplatin Phase 1: Pemetrexed (500, 600, 700, 800, or 900 mg/m^2) was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle.
  Carboplatin (AUC 5 or AUC 6 mg/mL*min) was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion.
  Participant accrual and dose escalations were dependent upon the observed pattern of dose limiting toxicity (DLT). If none of the 3 initial participants of a given dose level experienced a DLT in Cycle 1, enrollment proceeded to the next dose level.
Arm/Group | Pemetrexed/Carboplatin Phase 1
Number analyzed (Participants) | 0

2. Primary Outcome: Phase 2 - Percentage of Participants With Overall Tumor Response (Response Rate)
Description: Response is defined as CR (Complete Response) or PR (Partial Response) per Response Evaluation Criteria in Solid Tumor (RECIST criteria). Possible evaluations include: CR: Disappearance of all target lesions. PR: At least a 30% decrease in the size of target lesions.
  Response rate (%) = (number of patients with CR+PR/number of patients in Phase 2)*100
Time Frame: baseline to measured progressive disease (PD) (up to 18 months)
Population: Protocol Qualified (PQ) population. This population includes all patients in the Phase 2 study who met the following requirements:
  Histologic diagnosis of ovarian or primary peritoneal cancer, no concurrent chemotherapy, treatment with at least 1 dose of pemetrexed or 1 dose of carboplatin, presence of measurable disease as defined by RECIST.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed/Carboplatin Phase 2
Number analyzed (Participants) | 61
percentage of participants | 32.8 [21.3 to 46.0]

3. Secondary Outcome: Phase 1 - Number of Dose-Limiting Toxicities (DLTs)
Description: The following toxicities were considered DLT: CTCAE Grade 4 neutropenia (absolute neutrophil count [ANC] <0.5 × 10^9/L lasting ≥7 days. Febrile neutropenia (ANC <1.0 × 10^9/L, fever 38.5°C, and no documented infection). CTCAE Grade 4 thrombocytopenia (platelets <25.0 × 10^9/L).
  Any hemorrhage with CTCAE Grade ≥3 thrombocytopenia (50.0 × 10^9/L). CTCAE Grade ≥3 nonhematologic toxicity (excluding nausea, vomiting, or CTCAE Grade 3 alanine transaminase (ALT) or aspartate aminotransferase (AST) that returned to baseline prior to next treatment).
  Treatment delay more than 1 week due to toxicity.
Time Frame: baseline through end of Phase 1 (up to 18 months)
Population: Intention to Treat (ITT) population - all patients that consented and were successfully screened (note patient may or may not have received treatment; patients that were screen failures were not included in this population).
Measure: Number; unit: DLT events
Arm/Group | Pemetrexed/Carboplatin Phase 1
Number analyzed (Participants) | 20
DLT events
  Number of DLT Events | 1
  DLT Event: Grade 4 Neutropenia | 1

4. Secondary Outcome: Phase 1 - Number of Participants With Adverse Events (Toxicity)
Description: A listing of adverse events is located in the Reported Adverse Event module.
Time Frame: baseline measured to progressive disease (up to 18 months)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Pemetrexed/Carboplatin Phase 1
Number analyzed (Participants) | 20
Participants
  Serious Adverse Events | 2
  Other Adverse Events | 19

5. Secondary Outcome: Phase 1 - Recommended Dose of Pemetrexed for Phase 2
Description: MTD was to be used as Phase 2 recommended dose. MTD was to be determined by increasing doses of pemetrexed up to 900 mg/m^2 based on observed pattern of dose limiting toxicity (DLT: See Outcome #3). If none of 3 initial participants at a given level had a DLT in Cycle 1, enrollment proceeded to next dose level. If at least 2 participants had a DLT in Cycle 1 at a dose level, that dose level was considered the MTD. However, based on results from another Phase 2 Study (NCT00109096), further dose escalations were not explored and dose was selected based on results of that Phase 2 Study.
Time Frame: baseline measured to progressive disease (up to 18 months)
Population: as for outcome 3
Measure: Number; unit: mg/m^2 (milligrams per square meter)
Arm/Group | Pemetrexed/Carboplatin Phase 1
Number analyzed (Participants) | 20
mg/m^2 (milligrams per square meter) | 500

6. Secondary Outcome: Phase 1 - Recommended Area Under the Curve (AUC) Dose of Carboplatin for Phase 2
Description: MTD was to be used as Phase 2 recommended dose. MTD determined by increasing doses up to AUC 6 mg/mL*min based on pattern of DLT (Outcome #3). If none of 3 initial participants at given level had DLT in Cycle 1, enrollment proceeded to next dose level. If at least 2 participants had DLT in Cycle 1 at dose level, that dose level was considered MTD. However, based on results from Phase 2 Study (NCT00109096), further dose escalations were not explored: carboplatin dose was selected based on standard dose employed in control arm of first-line therapy for epithelial ovarian cancer (Bookman 2006).
Time Frame: baseline measured to progressive disease (up to 18 months)
Population: as for outcome 3
Measure: Number; unit: mg/mL*min
Arm/Group | Pemetrexed/Carboplatin Phase 1
Number analyzed (Participants) | 20
mg/mL*min | 6

7. Secondary Outcome: Phase 1 - Number of Participants With Tumor Response
Description: Patients were analyzed by Cancer Antigen-125 (CA-125) response criteria and RECIST guidelines. Possible evaluations include: Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the size of target lesions. Progressive Disease (PD): At least a 20% increase in the size of target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: baseline measured to progressive disease (up to 18 months)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Pemetrexed/Carboplatin Phase 1
Number analyzed (Participants) | 20
Participants
  Complete Response (CR) | 12
  Partial Response (PR) | 4
  Stable Disease (SD) | 1
  Progressive Disease (PD) | 2

8. Secondary Outcome: Phase 2 - Time to Response (TTR)
Description: Response is defined as CR (Complete Response) or PR (Partial Response) per RECIST criteria. Possible evaluations include: Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the size of target lesions. Progressive Disease (PD): At least a 20% increase in the size of target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: First treatment to response (up to 31 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Carboplatin Phase 2
Number analyzed (Participants) | 20
Months | 1.8 [1.4 to 2.8]

9. Secondary Outcome: Phase 2 - Duration of Response (DOR)
Description: Duration of response is defined as the time from first observation of Complete Response or Partial Response to the first observation of Progressive Disease or death from any cause. For patients who are still alive at the time of analysis, and who do not have Progressive Disease, duration of response will be censored at the date of the last objective progression-free disease assessment.
Time Frame: time of response to progressive disease (up to 31 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Carboplatin Phase 2
Number analyzed (Participants) | 20
Months | 9.1 [6.9 to 10.2]

10. Secondary Outcome: Phase 2 - Time to Disease Progression
Description: Time to objective progressive disease (TTPD) is defined as the time from the date of study enrollment to the date of objectively determined Progressive Disease (PD). For patients who die without objective PD (including death from study disease), TTPD will be censored at the date of the last objective progression-free disease assessment. For patients who are still alive at the time of analysis, and who do not have PD, TTPD will be censored at the date of the last objective progression-free disease assessment.
Time Frame: baseline to measured progressive disease (up to 31 months)
Population: Protocol Qualified (PQ) population. This population includes all patients in the Phase 2 study who met the following requirements:
  Histologic diagnosis of ovarian or primary peritoneal cancer, no concurrent chemotherapy, treatment with at least 1 dose of pemetrexed or 1 dose of carboplatin, presence of measurable disease as defined using RECIST.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Carboplatin Phase 2
Number analyzed (Participants) | 61
Months | 9.5 [8.3 to 11.3]

11. Secondary Outcome: Phase 2 - Time to Treatment Failure
Description: Time to treatment failure (TTTF) is defined as the time from the date of study enrollment to the date of the first observation of disease progression, death from any cause, or early discontinuation of treatment (any reason). For patients who are alive, progression-free, and have not discontinued early at the time of analysis, TTTF will be censored at the date of the last objective progression-free disease assessment.
Time Frame: First treatment to discontinuation of study drug, progressive disease, or death (up to 31 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Carboplatin Phase 2
Number analyzed (Participants) | 61
Months | 7.1 [4.6 to 8.5]

12. Secondary Outcome: Phase 2 - Overall Survival
Description: Overall survival is defined as the time from the date of study enrollment to the date of death from any cause. This analysis was not done due to the high number of censored patients.
Time Frame: baseline to date of death from any cause (up to 31 months)
Population: Protocol Qualified (PQ) population. This analysis was not done due to the high number of censored patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed/Carboplatin Phase 2
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase 2 - Number of Participants With Adverse Events (Toxicity)
Description: A listing of adverse events is located in the Reported Adverse Event module.
Time Frame: baseline through end of Phase 2 (up to 31 months)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Pemetrexed/Carboplatin Phase 2
Number analyzed (Participants) | 66
participants
  Serious Adverse Events | 15
  Other Adverse Events | 63

14. Secondary Outcome: Phase 2 - Progression-Free Survival
Description: Progression-free survival (PFS) is defined as the time from the date of study enrollment to the date of objectively determined PD or death from any cause, whichever comes first. For patients who are still alive at the time of analysis, and who do not have PD, PFS will be censored at the date of the last objective progression-free disease assessment.
Time Frame: baseline to measured progressive disease (up to 31 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Carboplatin Phase 2
Number analyzed (Participants) | 61
Months | 9.4 [8.3 to 11.1]

ADVERSE EVENTS:
Description: Adverse events are reported regardless of potential relatedness to study drug or Grade (severity).
Groups:
- Pemetrexed 500 + Carboplatin AUC 5 (Phase 1): Pemetrexed (500 mg/m^2) was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle. Carboplatin (AUC 5) was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion.
- Pemetrexed 600 + Carboplatin AUC 5 (Phase 1): Pemetrexed (600 mg/m^2) was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle. Carboplatin (AUC 5) was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion.
- Pemetrexed 600 + Carboplatin AUC 6 (Phase 1): Pemetrexed (600 mg/m^2) was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle. Carboplatin (AUC 6) was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion.
- Pemetrexed 700 + Carboplatin AUC 6 (Phase 1): Pemetrexed (700 mg/m^2) was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle. Carboplatin (AUC 6) was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion.
- Pemetrexed 800 + Carboplatin AUC 6 (Phase 1): Pemetrexed (800 mg/m^2) was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle. Carboplatin (AUC 6) was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion.
- Pemetrexed 900 + Carboplatin AUC 6 (Phase 1): Pemetrexed (900 mg/m^2) was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle.
  Carboplatin (AUC 6) was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion.
- Pemetrexed 500 + Carboplatin AUC 6 (Phase 2): Pemetrexed (500 mg/m^2) was administered intravenously over approximately 10 minutes on Day 1 of a 21-day cycle.
  Carboplatin (AUC 6) was administered intravenously over approximately 30 minutes on Day 1 of a 21-day cycle, beginning approximately 30 minutes after the end of the pemetrexed infusion.
Arm/Group | Pemetrexed 500 + Carboplatin AUC 5 (Phase 1) | Pemetrexed 600 + Carboplatin AUC 5 (Phase 1) | Pemetrexed 600 + Carboplatin AUC 6 (Phase 1) | Pemetrexed 700 + Carboplatin AUC 6 (Phase 1) | Pemetrexed 800 + Carboplatin AUC 6 (Phase 1) | Pemetrexed 900 + Carboplatin AUC 6 (Phase 1) | Pemetrexed 500 + Carboplatin AUC 6 (Phase 2)
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/4 | 0/3 | 1/3 | 1/3 | 15/66
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 3/3 | 3/3 | 2/3 | 63/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed 500 + Carboplatin AUC 5 (Phase 1) (N=4) | Pemetrexed 600 + Carboplatin AUC 5 (Phase 1) (N=3) | Pemetrexed 600 + Carboplatin AUC 6 (Phase 1) (N=4) | Pemetrexed 700 + Carboplatin AUC 6 (Phase 1) (N=3) | Pemetrexed 800 + Carboplatin AUC 6 (Phase 1) (N=3) | Pemetrexed 900 + Carboplatin AUC 6 (Phase 1) (N=3) | Pemetrexed 500 + Carboplatin AUC 6 (Phase 2) (N=66)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Zygomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed 500 + Carboplatin AUC 5 (Phase 1) (N=4) | Pemetrexed 600 + Carboplatin AUC 5 (Phase 1) (N=3) | Pemetrexed 600 + Carboplatin AUC 6 (Phase 1) (N=4) | Pemetrexed 700 + Carboplatin AUC 6 (Phase 1) (N=3) | Pemetrexed 800 + Carboplatin AUC 6 (Phase 1) (N=3) | Pemetrexed 900 + Carboplatin AUC 6 (Phase 1) (N=3) | Pemetrexed 500 + Carboplatin AUC 6 (Phase 2) (N=66)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 19 (32)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 2 (4) | 0 (0) | 20 (65)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 3 (3) | 1 (5) | 2 (3) | 0 (0) | 32 (109)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 3 (5) | 3 (3) | 2 (2) | 0 (0) | 14 (41)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratoconjunctivitis sicca (Eye disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 10 (19)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (7) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 9 (11)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (24) | 2 (12) | 2 (3) | 3 (9) | 1 (1) | 2 (4) | 21 (39)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 2 (5) | 0 (0) | 10 (16)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (6)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (15) | 2 (10) | 3 (9) | 3 (12) | 3 (12) | 2 (5) | 42 (108)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 10 (13)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (5) | 4 (8) | 3 (13) | 3 (8) | 1 (1) | 27 (45)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (15) | 2 (2) | 4 (7) | 2 (3) | 3 (5) | 1 (2) | 33 (57)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (18)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (8)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 17 (41)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (7)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (11)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (10)
Blood glucose increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 18 (27)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (44)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 16 (40)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (15)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 5 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Headache (Nervous system disorders) | 2 (4) | 3 (6) | 3 (6) | 1 (1) | 1 (1) | 2 (2) | 5 (10)
Neuropathy peripheral (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 6 (7)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 18 (19)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (3) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Leukoplakia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (10)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 10 (13)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 2 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (3) | 6 (12)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days